CLINICAL TRIAL: NCT03780933
Title: The Impact of High Dose Vitamin C "Ascorbic Acid" on the Clinical Outcomes of Critically Ill Patients With Acute Respiratory Distress Syndrome
Brief Title: the Effect of High Dose Ascorbic Acid on Critically Ill Patients With ARDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Misr International University (Other)
Responsible Party: Principal Investigator, Nada Hazem Farrag, Assistant Lecturer, Misr International University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 247
Record Dates: First submitted 2018-08-08; First posted 2018-12-19 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-10

CONDITIONS: Acute Respiratory Distress
MeSH Terms: conditions — Acute Lung Injury | interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): conventional treatment (corticosteroids, mechanical ventilation)
- test group (vitamin C) (Experimental): high dose vitamin c iv infusion
  Interventions: Dietary Supplement: vitamin c

INTERVENTIONS:
Dietary Supplement: vitamin c — vitamin c IV 10 G
  Arms: test group (vitamin C)

SUMMARY:
1. To access role of vitamin C supplementation in ARDS patients on the following:

   Oxidants/ antioxidants imbalance Length of hospital stay Mortality rate Weaning from mechanical ventilator Incidence of adverse drug reaction
2. To access tolerability of vitamin C supplementation in patients with ARDS.

DETAILED DESCRIPTION:
Acute Respiratory distress syndrome (ARDS) is a form of severe hypoxemic respiratory failure due to severe impairment of gas exchange and lung mechanics that is characterized by inflammatory injury to the alveolar capillary barrier, with extravasation of protein-rich edema fluid into the air space. Current ARDS antioxidant treatment strategy, is based upon supportive therapies including low tidal volume ventilation, fluid management, nutritional support and glucocorticoids.

Ascorbic acid or Vitamin C is an important dietary water-soluble antioxidant, it significantly decreases the adverse effects of ROS such as reactive oxygen and nitrogen species that can cause oxidative damage to macromolecules. Recent studies show that high dose of Vitamin C have protective effects against overwhelming oxidative stress due to critical illness. Vitamin C improves immune function and improves tissue perfusion and reduce tissue hypoxia and subsequent organ dysfunction. Also, Ascorbate, the redox form of vitamin C is physiological antioxidant and has bacteriostatic activity Hence the study aims to evaluate the impact of IV Vitamin C in ARDS, as a novel pharmaceutical approach in an attempt to improve the clinical outcome of ARDS patients, decrease other medications toxicities and improve patients' quality of life.

The objective of the current study was to evaluate the efficacy, safety and tolerability of IV Vitamin C administration in addition to conventional therapy in patients with ARDS by assessing the following:

1. Oxidants/ antioxidants imbalance
2. Length of hospital stay
3. Mortality rate
4. Weaning from mechanical ventilator
5. Incidence of adverse drug reaction
6. Serum IL8 levels

8. Serum Vitamin C levels

ELIGIBILITY:
Inclusion Criteria:

1. All ARDS cases presenting to the Chest department ICU within 48 hours of diagnosis
2. who don't have an exclusion criteria will be included.

Exclusion Criteria:

1. Known allergy to Vitamin C
2. Inability to obtain consent;
3. Age < 18 years;
4. More than 48 hours since meeting ARDS criteria;
5. Pregnancy or breast feeding,
6. Moribund patient not expected to survive 24 hours;
7. Patients not eligible to CPR
8. Active kidney stone

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2019-06-20 (Actual)

PRIMARY OUTCOMES:
Assessment of Improvement in ARDS patient's mortality rate | within 10 days of ARDS diagnosis
  Days to weaning from ventilator

SECONDARY OUTCOMES:
Intensive Care Unit Length of Stay | subject will be followed until discharged from the ICU, has deceased, or study duration has reached 10days from time of enrollment, whichever is first
  improvement in clinical outcome
Duration of Mechanical Ventilation | subject will be followed until mechanical ventilation has been discontinued, the subject has deceased, or study duration has reached 10 days from time of enrollment, whichever is first
  improvement in respiratory functions

CONTACTS AND LOCATIONS:
Overall Officials: Nada Farrag, Msc, Principal Investigator — Misr International University
Locations (1):
- Embaba Chest Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No